CLINICAL TRIAL: NCT04308226
Title: Lung Cancer Screening Navigation for Homeless People: A Pragmatic Trial
Brief Title: Lung Cancer Screening Navigation for Homeless People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Travis Paul Baggett, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2018P001344; RSG-17-157-01-CPPB (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer; Tobacco Use; Homelessness
Keywords: lung cancer screening; tobacco use; homeless persons; smoking; low-dose computed tomography
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use; Smoking | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to usual care with (N=200) or without (N=100) lung cancer screening (LCS) navigation. Randomization will be stratified by smoking status, housing status, clinical site, and whether participants have already discussed LCS with their primary care provider (PCP) to ensure balance between study arms on these variables.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care without patient navigation (No Intervention): Participants assigned to this arm will be given basic educational materials on general lung health and referred back to their primary care provider (PCP) for management as per usual practice.
- Usual care with patient navigation (Experimental): Participants assigned to this arm will be informed about lung cancer screening (LCS), provided educational materials on LCS and patient navigation, and offered access to an LCS navigator who will partner with participants and primary care providers (PCPs) to facilitate low-dose computed tomography (LDCT) completion and follow-up.
  Interventions: Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: Patient Navigation — The navigator's principal role is to guide participants through the lung cancer screening (LCS) process. The navigator will work within the existing Boston Health Care for the Homeless (BHCHP) clinical structure and collaborate with participants' primary care providers (PCPs) to facilitate LCS low-dose computed tomography (LDCT) referral, completion, and timely follow-up by addressing participants' barriers to LCS completion and enhancing participants' self-efficacy. The navigator's secondary role is to offer brief tobacco counseling for participants who currently smoke.
  Arms: Usual care with patient navigation

SUMMARY:
The investigators will conduct a pragmatic clinical trial to test the effect of patient navigation on lung cancer screening (LCS) low-dose computed tomography (LDCT) completion among Boston Health Care for the Homeless Program (BHCHP) patients at increased risk for lung cancer. Patient navigation is a strategy for guiding individuals through complex health systems, and the investigators hypothesize that this may be a promising approach for helping homeless-experienced people overcome their unique barriers to obtaining LCS.

The investigators will aim to recruit 300 people to participate in this research study; 100 will be randomly assigned to arm 1 (usual care) and 200 will be randomly assigned to arm 2 (patient navigation). Randomization of participants will be stratified by smoking status, housing status, clinical site, and whether they have previously discussed LCS with their primary care provider (PCP) to ensure balance between study groups on these variables. People assigned to the usual care arm will be referred back to their PCP for further management. People assigned to the patient navigation arm will be given the chance to work with a LCS navigator. The navigator will assist participants and their PCPs with all aspects of the LCS process in addition to offering brief tobacco counseling for current smokers.

The primary aim of the trial is to determine-among homeless-experienced people who are eligible for LCS-the effect of patient navigation on 1) LCS LDCT completion at 6 months post-enrollment and 2) LCS LDCT completion at 6 months with diagnostic follow-up of abnormal results within 1 month of the recommended time frame. Study outcomes will be assessed by examining participant health records.

Following the intervention, qualitative interviews will be conducted with 40 participants and 10 BHCHP PCPs to better understand how the LCS process unfolds in the setting of homelessness, the ways in which the navigator facilitated this process, and opportunities for improving the navigation intervention for future use.

ELIGIBILITY:
Inclusion Criteria:

* Currently or formerly homeless
* Have a 30 pack-year smoking history and have smoked within the past 15 years
* Have a Boston Health Care for the Homeless (BHCHP) primary care provider (PCP)
* Proficient in English, assessed with items asking about native language and self-reported comfort communicating in English among non-native speakers

Exclusion Criteria:

* Prior chest computed tomography (CT) imaging in the past 12 months
* Personal history of lung cancer, or current presentation with symptoms concerning for lung cancer (e.g. hemoptysis or unexplained weight loss of >15 lbs. in the past year)
* PCP is the principal investigator
* Inability to provide informed consent, assessed with knowledge questions about the material presented during the informed consent process that individuals must correctly answer before providing informed consent to participate

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Travis P Baggett, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Boston Health Care for the Homeless Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baggett TP, Sporn N, Barbosa Teixeira J, Rodriguez EC, Anandakugan N, Little BR, Chang Y, Park ER, Rigotti NA, Fine DR. Homelessness, Patient Navigation, and Lung Cancer Screening in a Health Center Setting: A Subgroup Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2519780. doi: 10.1001/jamanetworkopen.2025.19780. PMID 40674053
- [Derived] Baggett TP, Sporn N, Barbosa Teixeira J, Rodriguez EC, Anandakugan N, Critchley N, Kennedy E, Hart K, Joyce A, Chang Y, Percac-Lima S, Park ER, Rigotti NA. Patient Navigation for Lung Cancer Screening at a Health Care for the Homeless Program: A Randomized Clinical Trial. JAMA Intern Med. 2024 Aug 1;184(8):892-902. doi: 10.1001/jamainternmed.2024.1662. PMID 38856994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial recruitment occurred between 2020-2022. The trial was conducted at Boston Health Care for the Homeless Program (BHCHP), a federally-qualified healthcare for the homeless program that serves nearly 10,000 patients each year across more than 30 service sites in greater Boston (www.bhchp.org). Individuals were recruited through a combination of in-person and phone-based outreach as well as referrals from BHCHP primary care providers.
Pre-assignment Details: In total, 261 participants enrolled but one participant chose to withdraw before completing the baseline survey and therefore could not be randomized.
Period: Overall Study
Arm/Group | Usual Care Without Patient Navigation | Usual Care With Patient Navigation
Started | 87 | 173
Completed | 87 | 173
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Without Patient Navigation | Usual Care With Patient Navigation | Total
Number analyzed (Participants) | 87 | 173 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (5.4) | 60.5 (4.4) | 60.5 (4.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 61 | 123 | 184
  Female | 24 | 50 | 74
  Other | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — 4 participants had unknown race/ethnicity due to item non-response.
  Participants
    Hispanic/Latinx | 14 | 24 | 38
    Non-Hispanic Black | 30 | 66 | 96
    Non-Hispanic White | 29 | 67 | 96
    Non-Hispanic Other | 12 | 14 | 26
    Unknown | 2 | 2 | 4
Housing status [Count of Participants; unit: Participants] — Operationalization of current homelessness is concordant with the definition in the HEARTH Act of 20091 and used by the US Department of Housing and Urban Development.
  Participants
    Currently homeless | 28 | 56 | 84
    Formerly homeless | 59 | 117 | 176
Health insurance [Count of Participants; unit: Participants]
  With health insurance | 86 | 173 | 259
  Without health insurance | 1 | 0 | 1
Primary care location [Count of Participants; unit: Participants]
  BHCHP program headquarters | 63 | 121 | 184
  BHCHP satellite site | 24 | 52 | 76
Prior discussion of LCS with PCP [Count of Participants; unit: Participants] — Whether participants had ever discussed lung cancer screening with their primary care provider prior to study enrollment (self-reported).
  Participants
    Yes | 32 | 67 | 99
    No | 55 | 106 | 161
General self-efficacy score [Mean (Standard Deviation); unit: units on a scale] — Score range 10-40; higher scores represent greater self-efficacy.
  units on a scale | 32.4 (5.2) | 32.6 (5.8) | 32.5 (5.6)
Health status [Count of Participants; unit: Participants] — Based on a single-item assessment of self-rated health.
  Participants
    Fair/poor | 46 | 86 | 132
    Excellent/very good/good | 41 | 87 | 128
Mental health problem [Count of Participants; unit: Participants] — Defined as a score ≥13 on the 6-item Kessler Psychological Distress Scale (K6); 2 participants with status unknown due to item non-response.
  Participants
    Yes | 24 | 51 | 75
    No | 62 | 121 | 183
    Unknown | 1 | 1 | 2
Alcohol use problem [Count of Participants; unit: Participants] — Defined as a score ≥3 on the Alcohol Use Disorders Identification Test - Concise (AUDIT-C); 5 participants with status unknown due to item non-response.
  Participants
    Yes | 16 | 45 | 61
    No | 68 | 126 | 194
    Unknown | 3 | 2 | 5
Drug use problem [Count of Participants; unit: Participants] — Defined as a score ≥3 on the Drug Abuse Screening Test (DAST-10); 1 participant with status unknown due to item non-response.
  Participants
    Yes | 21 | 51 | 72
    No | 65 | 122 | 187
    Unknown | 1 | 0 | 1
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 75 | 146 | 221
  Former smoker | 12 | 27 | 39
Pack-years of smoking [Mean (Standard Deviation); unit: pack-years] — Calculated by multiplying the number of years of smoking by the typical number of packs per day consumed during those years.
  pack-years | 50.1 (21.5) | 47.1 (18.3) | 48.1 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Number (Percentage) of Participants Who Receive Low-dose Computed Tomography (LDCT) for Lung Cancer Screening (LCS) at 6 Months (26 Weeks).
Description: This outcome will be based on radiology records verifying that a chest computed tomography (CT) was performed for LCS and interpreted according to the lung imaging reporting and data system (Lung-RADS) framework.
Time Frame: 6 months (26 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Without Patient Navigation | Usual Care With Patient Navigation
Number analyzed (Participants) | 87 | 173
Participants | 8 | 75
Statistical Analysis 1: Comparison: Usual Care Without Patient Navigation vs Usual Care With Patient Navigation; Test type: Superiority; p < 0.001, Chi-squared

2. Secondary Outcome: Number (Percentage) of Participants Who Receive Low-dose Computed Tomography (LDCT) for Lung Cancer Screening (LCS) at 6 Months (26 Weeks) With Diagnostic Follow-up of Abnormal Results Within 1 Month (4 Weeks) of the Recommended Time Frame.
Description: Participants must achieve the primary outcome and, if the result is abnormal (lung imaging reporting and data system lung imaging reporting and data system (Lung-RADS) category 3 or 4), also obtain the next recommended follow-up test within 1 month (4 weeks) of the advised timeframe based on the Lung-RADS framework. Radiology records will be obtained for participants who underwent LDCT for LCS to document the findings of the study, determine the Lung-RADS category associated with those findings, and ascertain the recommended diagnostic follow-up plan.
Time Frame: 6 months (26 weeks) plus guideline-recommended follow-up timeframe plus 1 month (4 weeks)
Population: Participants who completed LDCT for LCS with Lung-RADS scores ≥3 meriting earlier than annual follow-up (typically 6 months for Lung-RADS 3, 3 months for Lung-RADS 4A, and immediate for Lung-RADS 4B/X). In the usual care without patient navigation arm, 1 participant received a Lung-RADS score of 4A. In the usual care with patient navigation arm, 6 participants received a Lung-RADS score of 3, 2 participants received a score of 4A, and 1 participant received a score of 4B.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Without Patient Navigation | Usual Care With Patient Navigation
Number analyzed (Participants) | 1 | 9
Participants | 1 | 2

3. Other Pre Specified Outcome: Time to Completion of Low-dose Computed Tomography (LDCT) for Lung Cancer Screening (LCS)
Description: Time between date of randomization and date of receipt of low-dose computed tomography (LDCT) for lung cancer screening (LCS) or date of censoring (6 months / 26 weeks)
Time Frame: 6 months (26 weeks)
Population: Outcome summarized by 25th percentile achieving completion.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Usual Care Without Patient Navigation | Usual Care With Patient Navigation
Number analyzed (Participants) | 87 | 173
weeks | NA [NA to NA] — "Median" is used here to indicate 25th percentile. Not enough participants in this arm achieved the outcome to calculate the 25th percentile and 95% confidence interval. | 9.7 [7.3 to 12.1]
Statistical Analysis 1: Comparison: Usual Care Without Patient Navigation vs Usual Care With Patient Navigation; Test type: Superiority; p < 0.001, Log Rank

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care Without Patient Navigation | Usual Care With Patient Navigation
All-Cause Mortality (participants affected / at risk) | 1/87 | 1/173
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/173
Other Adverse Events (participants affected / at risk) | 0/87 | 0/173

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04308226/Prot_SAP_000.pdf